CLINICAL TRIAL: NCT01506557
Title: Effect of Vitamin D Supplementation During Lactation on Vitamin D Status, Bone Mineralisation and Body Composition of Mother and Their Exclusively Breastfed Infants.
Brief Title: Vitamin D Supplementation of Lactating Mothers
Acronym: MAVID
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Children's Memorial Health Institute, Poland (Other)
Collaborators: Nutricia Research Fundation (Other)
Responsible Party: Principal Investigator, Justyna Czech-Kowalska, Deputy Head of Neonatology and Intensive Care, MD, PhD, Children's Memorial Health Institute, Poland
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 763/10
Record Dates: First submitted 2011-05-11; First posted 2012-01-10 (Estimated); Last update posted 2013-07-23 (Estimated); Status verified 2013-07

CONDITIONS: Vitamin D Deficiency
Keywords: vitamin D; vitamin D deficiency; breastfeeding; body composition; bone mineral content
MeSH Terms: conditions — Vitamin D Deficiency; Breast Feeding | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- choecalciferol (Experimental)
  Interventions: Dietary Supplement: cholecalciferol
- placebo (Placebo Comparator)
  Interventions: Dietary Supplement: placebo

INTERVENTIONS:
Dietary Supplement: cholecalciferol — dose 800 IU/day for 6 month
  Other Names: vit D
  Arms: choecalciferol
Dietary Supplement: placebo — oil capsules
  Arms: placebo

SUMMARY:
The investigators would like to test the hypothesis that maternal vitamin D supplementation during lactation in dose 1200IU/d (400IU from multivitamins + 800 IU cholecalciferol) is more effective than 400IU/d (400IU from multivitamins + placebo)to built appropriate maternal vitamin D status and could be beneficial for maternal and infants bone mineralization and body composition (proper proportion of muscle and fat tissues in body weight) and is safe for both.

The investigators also want to confirm that vitamin D supplementation of exclusively breastfed infants in dose 400IU/d is adequate to build appropriate vitamin D status independently of mother's vitamin D supplementation up to 1200 ID/d.

Additionally the investigators hypothesize that because of changes in lifestyle there will be no substantial seasonal differences in vitamin D status of pregnant women at the delivery and their newborn infants.

ELIGIBILITY:
Inclusion Criteria:

* Healthy women without major medical problem delivered at term and planning breastfeeding for next six months delivering term, single, infants with birth weight appropriate for gestational age without major health problem

Exclusion Criteria:

* Maternal endocrine disorders, disturbed calcium- phosphorus homeostasis, anticonvulsant treatment.
* Infants renal, hepatic insufficiency, endocrine disorders, congenital malformations, anticonvulsant treatment.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 174 (Actual)
Dates: Start 2011-03; Primary Completion 2012-10 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
serum 25-hydroxyvitamin D concentration, | 3 time poits up to 6 months (0-3-6 months)

SECONDARY OUTCOMES:
body composition measured by dual x-ray densitometry | 3 time points up to 6 months (0-3-6months)
serum calcium | 2 time poits up to 6 months ( 3-6 months)
calciuria (Urinary calcium and creatinine - UCa/crea) | 2 time poits up to 6 months ( 3-6 months)
iPTH | 3 time poits up to 6 months (0-3-6 months)
Prevalence of vitamin D deficiency (25OHD<20ng/ml) | 3 time poits up to 6 months (0-3-6 months)
Prevalence of vitamin D sufficiency (25OHD>30ng/ml) | 3 time poits up to 6 months (0-3-6 months)

CONTACTS AND LOCATIONS:
Overall Officials: Justyna Czech-Kowalska, MD, PhD, Principal Investigator — The Children's Memorial Health Institute
Locations (5):
- Poland (5):
  - Public Hospital, Otwock, Warsaw
  - Anna Mazowiecka Hospital, Warsaw Medical University, Warsaw
  - Gynecological and Obstetric Hospital, Warsaw
  - The Children's Memorial Health Institute, Warsaw
  - Międzyleski Hospital,, Warsaw

REFERENCES:
- [Derived] Czech-Kowalska J, Latka-Grot J, Bulsiewicz D, Jaworski M, Pludowski P, Wygledowska G, Chazan B, Pawlus B, Zochowska A, Borszewska-Kornacka MK, Karczmarewicz E, Czekuc-Kryskiewicz E, Dobrzanska A. Impact of vitamin D supplementation during lactation on vitamin D status and body composition of mother-infant pairs: a MAVID randomized controlled trial. PLoS One. 2014 Sep 18;9(9):e107708. doi: 10.1371/journal.pone.0107708. eCollection 2014. PMID 25232839